CLINICAL TRIAL: NCT05176977
Title: Using Data Analytics and Targeted Whole Health Coaching to Reduce Frequent Utilization of Acute Care Among Homeless Veterans
Brief Title: Homeless Veterans and Peer Whole Health Coaching
Acronym: PWHC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 19-187
Record Dates: First submitted 2021-12-16; First posted 2022-01-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Care Service Utilization; Mental Health Status; Physical Health Status; Housing
Keywords: Homeless Persons; Costs and Cost Analysis; Mental Health; Peer Support
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer Specialist - Whole Health Coaching (PS-WHC) (Experimental): Participants will meet with a Peer Specialist for 18 sessions over 24 weeks. The essential elements of this intervention include 1) general support provided via the core functions of a Peer Specialist, and 2) a structured Whole Health Coaching curriculum.
  Interventions: Behavioral: Peer Support-Whole Health Coaching
- Enhanced Usual Care (EUC) (No Intervention): Usual PACT care plus Hot Spotter Analytics (consists of access to field-based dashboard that allows PACTS to identify homeless Veterans on their panels who were super-utilizers, and the hot spotter manual).

INTERVENTIONS:
Behavioral: Peer Support-Whole Health Coaching — Participants will meet with a Peer Specialist for 18 sessions over a period of 24 weeks. The essential elements of this intervention include 1) general support provided via the core functions of a Peer Specialist and 2) a structured Whole Health Coaching curriculum.
  Other Names: PS-WHC
  Arms: Peer Specialist - Whole Health Coaching (PS-WHC)

SUMMARY:
Use of acute care services (e.g., hospitalizations, Emergency Department visits) contributes substantially to the cost of healthcare for Veterans. Homelessness is a robust social determinant of super utilization of acute care. The goal of this project is to test if Peer Specialists trained in Whole Health Coaching can reduce homeless Veterans' frequent use of acute care.

DETAILED DESCRIPTION:
Ten percent of patients account for up to 70% of acute care costs. Among these "super-utilizer" patients, homelessness is a robust social determinant of acute care utilization. Through a field-based dashboard and clinical aids, the Hot Spotter Analytic program assists Patient Aligned Care Teams (PACT) with targeting and tailoring care for the highest-need homeless Veterans. However, many Veterans identified by the Analytics do not engage in supportive services that reduce risk for acute care utilization. Peer Specialists (PS) are a high-value workforce that can facilitate Veterans' engagement in care. Yet, there is a need to enhance the PS role with a structured approach that can capitalize on known facilitators of care engagement among homeless Veterans. Whole Health Coaching (WHC) is one such approach. By focusing on patients' values and goals rather than treatment of specific conditions, WHC reduces patients' stigma regarding their care needs and increases patient activation and well-being, which can increase engagement in supportive services.

The goal of this project is to integrate use of Hot Spotter Analytics with Peer Specialists trained in Whole Health Coaching (PS-WHC) and evaluate whether this approach reduces homeless Veterans' frequent use of acute care. Using a Hybrid Type 1 design at the Palo Alto, Bedford, and North Little Rock VAs, the investigators will test whether receipt of PS-WHC (vs. Enhanced Usual Care; EUC) predicts (1a) lower acute care utilization, (1b) better health-related outcomes, and whether (1c) the effects of PS-WHC on 1a and 1b are mediated by increased (i) patient activation and well-being, and (ii) access to supportive services. Aim 2: Conduct a process evaluation to inform VA's potential widespread implementation of Hot Spotter Analytics + PS-WHC on PACTs. Aim 3: Conduct a Budget Impact Analysis to determine the impact on total costs of VA care due to implementing PS-WHC.

ELIGIBILITY:
Inclusion Criteria:

Veterans who:

* are on VA's Homeless Registry, which comprises those who utilized any VA homeless programs and services in the past 2 years
* are enrolled on a Patient Aligned Care Team (or "PACT") at a study site
* had a hot spotter qualifying event in two or more quarters in the past year will be eligible for participation

Exclusion Criteria:

* Veterans who have a suicidal and/or behavioral flag in their medical record and those who are too cognitively impaired to understand the informed consent process and other study procedures will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Days of all-cause hospitalization | 9 months (post-baseline)
  Data on all-cause hospitalization (medical/surgical, substance use, and mental health) (bed days of care) will be obtained from the CDW Inpatient and Outpatient files. VA-paid acute care at non-VA facilities will also be searched in the Fee Basis and Program Integrity Tool (PIT) files, including "Choice" care.

SECONDARY OUTCOMES:
ED visits | 9 months (post-baseline)
  Data on ED visits will be obtained from the CDW Inpatient and Outpatient files. VA-paid acute care at non-VA facilities will also be searched in the Fee Basis and Program Integrity Tool (PIT) files, including "Choice" care.
Substance Use | 9 months (post-baseline)
  The WHO-ASSIST measure will provide information on quantity and frequency of substance use, separately by drug type, in the past 30 days at each follow-up assessment.
Alcohol Use Problems (AUDIT) | 9 months (post-baseline)
  The AUDIT is an alcohol screen that help identify patients who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). Each of the 10 items on this scale has response options from 0 to 4; scores on the outcome measure can range from 0 to 40 with higher scores indicating more alcohol use problems.
Depression (PHQ-9) | 9 months (post-baseline)
  The Patient Health Questionnaire-9 (PHQ-9) will obtain information on changes in depression symptoms over time. The scale consists of 9 items, each answered on 4-point scale (0=not at all, 4=nearly every day). Scores on this outcome measure can range from 0 to 27, with higher scores indicating more symptoms of depression.
PTSD (PCL-5) | 9 months (post-baseline)
  The PTSD Checklist (PCL-5) will obtain information on changes in PTSD symptoms over time. The scale consists of 20 items, each answered on a 5-point scale (0=not at all, 4=extremely). Scores on the outcome measure can range from 0 to 80 with higher scores indicating more symptoms of PTSD.
Days of Ambulatory Care Sensitive Condition (ACSC) hospitalizations | 9 months (post-baseline)
  Ambulatory Care Sensitive Conditions (ACSCs) are a set of conditions such as asthma and diabetes, where the need for emergency admissions is thought to be avoidable. We will use the Agency for Healthcare Research and Quality (AHRQ)'s definition of the Prevention Quality Indicators (PQIs) as our definition of hospitalizations for ACSC. Data on ACSC hospitalizations will be obtained from the CDW Inpatient and Outpatient files. VA-paid acute care at non-VA facilities will also be searched in the Fee Basis and Program Integrity Tool (PIT) files, including "Choice" care.
Percent Days Homeless | 9 months (post-baseline)
  The reliable and valid Residential Timeline Followback (TLFB) interview will measure duration and frequency of homelessness (e.g., percent days homeless) in the past 90 days at baseline and each follow-up.
Days of mental health hospitalizations | 9 months (post-baseline)
  Data on mental health hospitalizations, including for substance use, will be obtained from the CDW Inpatient and Outpatient files. VA-paid acute care at non-VA facilities will also be searched in the Fee Basis and Program Integrity Tool (PIT) files, including "Choice" care.
Patient Engagement (ACE) | 9 months (post-baseline)
  The 21-item Altarum Consumer Engagement (ACE) Measure is a reliable and valid self-report measure of patient activation, which yields a total score. Items are answered on a 5-point scale (0=strongly disagree, 4=strongly agree). A total score is calculated ranging from 0 to 100, with higher scores indicating greater patient engagement/activation in their health care.
Days of medical hospitalizations | 9 months (post-baseline)
  Data on medical hospitalizations will be obtained from the CDW Inpatient and Outpatient files. VA-paid acute care at non-VA facilities will also be searched in the Fee Basis and Program Integrity Tool (PIT) files, including "Choice" care.
Perceptions of Health (PROMIS-10) | 9 months (post-baseline)
  Global health items from the Patient Reported Outcome Measurement Information System (PROMIS) will assess perceptions of health. Comprised of 10 items, this measure will assess participants' perception of their overall health and quality of life, as well as their physical, mental, and social health. Scores
Peer service engagement | 9 months (post-baseline)
  Data on peer services (number of encounters) will be obtained from the CDW Inpatient and Outpatient files.
Whole Health service engagement | 9 months (post-baseline)
  Data on Whole Health services, including Complementary and Integrative Health (CIH) services, (number of encounters) will be obtained from the CDW Inpatient and Outpatient files.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Blonigen, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA; David A. Smelson, PsyD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (3):
- United States (3):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blonigen D, Hyde J, McInnes DK, Yoon J, Byrne T, Ngo T, Smelson D. Integrating data analytics, peer support, and whole health coaching to improve the health outcomes of homeless veterans: Study protocol for an effectiveness-implementation trial. Contemp Clin Trials. 2023 Feb;125:107065. doi: 10.1016/j.cct.2022.107065. Epub 2022 Dec 23. PMID 36572239

DOCUMENTS (1):
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT05176977/ICF_000.pdf